CLINICAL TRIAL: NCT01429090
Title: Bioavailability of Vagantin® Coated Tablets Relative to an Oral Methantheline Bromide Solution
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: RIEMSER Arzneimittel GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BAMB0199
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-09

CONDITIONS: Neurogenic Bladder
Keywords: Pharmacokinetics; Accommodation, Ocular; Reflex, Pupillary; Salivation
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Sialorrhea | interventions — Blood Specimen Collection; Methantheline

ARMS (2):
- Test (Experimental): Pharmacokinetics and -dynamics after single dose administration of 2 coated tablets Vagantin® (coated tablets of 50 mg methantheline bromide)
  Interventions: Procedure: blood sampling; Drug: Vagantin®; Procedure: Measurement of salivation; Procedure: Measurement of accommodation; Procedure: Pupillometry
- Reference (Active Comparator): Pharmacokinetics and -dynamics after single dose administration 100 ml methantheline solution (100 mg methantheline bromide)
  Interventions: Procedure: blood sampling; Drug: methantheline solution; Procedure: Measurement of salivation; Procedure: Measurement of accommodation; Procedure: Pupillometry

INTERVENTIONS:
Procedure: blood sampling — blood sampling before and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 16 hours after administration of study medication
Drug: Vagantin® — administration of 2 coated tablets Vagantin® (coated tablets of 50 mg methantheline bromide)
  Arms: Test
Drug: methantheline solution — administration 100 ml methantheline solution (100 mg methantheline bromide)
  Arms: Reference
Procedure: Measurement of salivation — Volume of salivary gland secretion was measured by chewing a 5 x 5 cm piece of PARAFILM "M"® (American Can Company, UK) for 5 min. Saliva was collected in glass tubes and the amount of the stimulated saliva was measured by weighing
Procedure: Measurement of accommodation — Accommodation was measured with the optometer according to Schober (Velhagen 1972)
Procedure: Pupillometry — Pupil function was assessed with the pupillograph (Compact Integrated Pupillograph, AMTech, Weinheim, Germany). The following data were obtained: pupil diameter, response to defined flash stimuli

SUMMARY:
The primary objective of the study is:

•To describe extent and rate of absorption of methantheline after single oral dose administration of Vagantin® coated tablets (Test) in comparison to a methantheline bromide solution (Reference)

The secondary objectives of the study are:

* To determine elimination the half-life of methantheline bromide
* To describe the effects of Test and Reference on salivation, accommodation, pupil response, blood pressure and heart rate
* to assess frequency and intensity of adverse drug reactions

DETAILED DESCRIPTION:
The quarternary anticholinergic compound methantheline bromide (diethyl-methyl [2-(9 xanthenyl carbonyloxy) ethyl] ammonium bromide) is marketed to treat neurogenic bladder instability. In comparison with atropine, it influences the parasympathetic nervous transmission more by ganglionic rather than peripheral muscarinic receptor blockade. Clinical effects after single therapeutic doses of 50-100 mg last for about 6 hours which is longer than after atropine. The drug relaxes smooth muscles of the gastrointestinal and urogenital tract. Furthermore, it inhibits bronchial, salivary and sweat glands secretion, lowers the production of gastric juice and disturbs accommodation.

There are no data available on the pharmacokinetic properties of methantheline in man. However, 25-50 mg intravenous methantheline seem to be equivalent to 50-100 mg p.o. with regard to the pharmacodynamic effects [Stille 1988].

Vagantin® is marketed as coated tablets containing 50 mg methantheline bromide. Because of the particular properties of methantheline (narrow therapeutic range, obviously erratic, incomplete and irregular absorption) and because of the national and international recommendations concerning the registration of drugs, Vagantin® must be evaluated with regard to its pharmacokinetic properties at least relative to a non-formulated form.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 - 45 years
* sex: male and female
* ethnic origin: Caucasian
* body weight: ±20 % of normal weight (Broca)
* good health as evidenced by the results of the clinical examination and the laboratory check-up which are judged by the clinical investigator not to differ in a clinical relevant way from the normal state
* written informed consent

Exclusion Criteria:

* known hypersensitivity to the investigational products or to their adjuvants
* pollakisurie of cardial and renal reasons
* megacolon
* atonia of the gastrointestinal tract
* atonia or hypotonia of the urinary bladder
* tachycardiac arrhythmia
* subvesical bladder obstruction, especially benign prostatic hypertrophy
* narrow angle glaucoma
* glasses or contact lenses
* history of gastrointestinal diseases (except appendectomy)
* history of renal and/or hepatic diseases
* any disease known to modify absorption, metabolism or excretion of the drug under investigation
* liability to orthostatic dysregulation, faintings, or blackouts
* alcohol consumption more than 40 g/day
* smokers of more than 10 cigarettes per day
* special or uniform nutritional habits, e.g. vegetarians or under-caloric diet
* less than 14 days after last acute disease
* less than 14 days after last systemic or local drug administration or 10 times the half life of the respective drug (except hormonal contraceptives)
* blood donation within the last two months
* blocking period due to another clinical study with investigational products; however at least 4 weeks after the end of the study or 10 times the half life of the respective drug
* lack of willingness or inability to co-operate adequately
* HIV and HBV and drug screening positive or not performed (in case of a positive HIV-test, the volunteers must be informed by a physician in a personal conversation)
* lactation and pregnancy test positive or not performed

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 1999-10; Primary Completion 1999-11 (Actual); Study Completion 2000-01 (Actual)

PRIMARY OUTCOMES:
area under the curve (AUC0-∞) | 0-16 h plasma concentration-time profile of methantheline after single oral administration
  AUC0-∞ was assessed by the trapezoidal formula up to the last sampling time with a concentration above the limit of quantitation (AUC0-), and was extrapolated to infinity using standard techniques
maximal plasma concentration (Cmax) | 0-16 h plasma concentration-time profile of methantheline after single oral administration
  Cmax was obtained directly from the measured concentration-time curves

SECONDARY OUTCOMES:
time of maximal plasma concentration (tmax) | 0-16 h plasma concentration-time profile of methantheline after single oral administration
  tmax was obtained directly from the measured concentration-time curves
terminal half-life (t½) | 0-16 h plasma concentration-time profile of methantheline after single oral administration
  Half-life (t½) was evaluated by non-linear regression of the terminal slope
volume of salivary gland secretion | before and 0, 0.5, 1, 2, 3, 4, 6, 8, 12 hours after administration of study medication
  Volume of salivary gland secretion will be measured by chewing a 5 x 5 cm piece of PARAFILM "M"® (American Can Company, UK) for 5 min. Saliva will be collected in glass tubes the volume of which will be measured be weighing
Measurement of accommodation | before and 0, 1, 2, 3, 4, 6, 8, 12 hours after administration of study medication
  Accommodation will be measured with the optometer according to Schober (Velhagen 1972)
Pupil function | before and 0, 1, 2, 3, 4, 6, 8, 12 hours after administration of study medication
  Pupil function will be assessed with the pupillograph (Compact Integrated Pupillograph, AMTech, Weinheim, Germany). The following data will be obtained: pupil diameter, response to defined flash stimuli

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology at the University of Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany

REFERENCES:
- [Derived] Muller C, Lotsch J, Giessmann T, Franke G, Walter R, Zschiesche M, Siegmund W. Relative bioavailability and pharmacodynamic effects of methantheline compared with atropine in healthy subjects. Eur J Clin Pharmacol. 2012 Nov;68(11):1473-81. doi: 10.1007/s00228-012-1286-6. Epub 2012 Apr 21. PMID 22527350